CLINICAL TRIAL: NCT04936412
Title: Clinical Comparative Study of Personalized Shoulder, Knee and Ankle Brace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jia-kuo yu (Other)
Responsible Party: Sponsor-Investigator, Jia-kuo yu, Peking University Third Hospital, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Personalized brace
Record Dates: First submitted 2018-05-27; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Shoulder Injuries; Knee Injuries; Ankle Injuries
Keywords: Personalized; brace; shoulder; knee; ankle
MeSH Terms: conditions — Shoulder Injuries; Knee Injuries; Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized brace group (Experimental): Personalized brace for patients
  Interventions: Device: Rehabilitation brace
- Conventional brace group (Active Comparator): Conventional brace for patients
  Interventions: Device: Rehabilitation brace

INTERVENTIONS:
Device: Rehabilitation brace — Rehabilitation brace
  Other Names: Individualized rehabilitation support

SUMMARY:
This study is based on human anatomical data and uses computer-aided engineering (CAE) software such as biomedical image processing software, reverse engineering software, CAD software, and finite element analysis software to create a three-dimensional bracing model. With the help of 3D printing technology, we have developed personalized brace, completed the personalized rapid design and optimization of the three series of support equipment products such as the posterior cruciate ligament brace, ankle ankle brace, and shoulder brace.

DETAILED DESCRIPTION:
The traditional brace mainly includes small splints or gypsums. The manufacturing process is rough, and the flexibility is poor. In recent years, with the development of orthopedic surgery, rehabilitation concept, modern polymer materials, and biomechanics, great progress has been made in R&D, production, and assembly of orthoses. In developed countries, orthoses is not only widely used after orthopedic surgery and the department of rehabilitation, but it has become the main auxiliary device for sports trauma surgery, immobilization, treatment, and rehabilitation training. Leading bracing company such as DJO has developed multi-brand correction devices such as Aircast®, Chattanooga, CMF, COMPEX®, DonJoy®, Empi® and ProCare®. However, these braces are not designed and manufactured based on patients. Individually designed products for anatomical structures still have many problems in clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* patients accepting arthroscopic surgery of the shoulder, posterior cruciate ligament reconstruction surgery, Achilles tendon rupture repair surgery.

Exclusion Criteria:

* Severe peripheral ligament injury of should, knee and ankle.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
appearance score | six weeks after injury
  Patient's preference for appearance
comfort score | two weeks after injury
  Patient comfort score
Convenience score | six weeks after injury
  Convenience of adjustment during rehabilitation
Satisfaction score | six weeks after injury
  Overall satisfaction of patients

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lin, Study Director — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No